CLINICAL TRIAL: NCT06368063
Title: Study on the Efficacy and Safety of Huaier Granule in Postoperative Adjuvant Therapy of Resectable Pancreatic Cancer
Brief Title: The Study of Huaier Granule in Postoperative Adjuvant Therapy of Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zheng Wang, professor, Xi'an Jiaotong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202301
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer Resectable
Keywords: Huaier granule; Postoperative adjuvant therapy; Resectable pancreatic cancer; Efficacy and safety
MeSH Terms: interventions — Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier treatment group (Experimental): The subjects take Huaier granules orally and start taking them within 15-30 days after surgery until the end of the study, intolerable toxicity occurs, withdrawal from the study for any reason, or death, whichever occurs first; Or the researcher determines that the subjects no longer benefit.
  Interventions: Drug: Huaier granule
- Standard chemotherapy group (Active Comparator): Accept treatment with Class 1A chemotherapy drugs recommended by CSCO (choose any one to receive treatment)
  * Gemcitabine combine with capecitabine
  * mFOLFIRINOX solution
  * Gemcitabine monotherapy
  * Tegafur，gimeracil and oteracil potassium capsules monotherapy
  Interventions: Drug: chemotherapy drugs

INTERVENTIONS:
Drug: Huaier granule — Huaier Granules: Oral administration, 10g once, 3 times a day, starting from 15-30 days after surgery until the end of the study, intolerable toxicity, withdrawal from the study for any reason, or death, whichever occurs first; Or the researcher determines that the subjects no longer benefit.
  Other Names: Z20000109#NMPA Approval Number#
  Arms: Huaier treatment group
Drug: chemotherapy drugs — Accept treatment with Class 1A chemotherapy drugs recommended by CSCO (choose any one to receive treatment)
  · Gemcitabine combine with capecitabine
  Gemcitabine 1000mg/m^2 intravenous infusion for more than 30 minutes, day 1, 8, 15,repeat every 4 weeks for a total of 6 cycles.
  · mFOLFIRINOX solution
  Oxaliplatin 85mg/m^2 intravenous infusion for 2 hours, day 1 Ilitacan 150mg/m^2 intravenous infusion for more than 30-90 minutes, day 1 Leucovorin calcium 400mg/m^2 intravenous infusion for 2 hours, day 1 5-FU 2400mg/m^2, continuous intravenous infusion for 46 hours, repeated every 2 weeks, administered until 24 weeks.
  * Gemcitabine monotherapy
    1000mg/m^2 intravenous infusion, day 1 qw x 7, rest for 1 week Afterwards, qw × 3, take a week off, and administer medication for 6 months.
  * Tegio capsules monotherapy
  Take tegio capsules orally, 80mg/d, day 1-28, repeated every 6 weeks, administered until 6 months.
  Other Names: Standard chemotherapy
  Arms: Standard chemotherapy group

SUMMARY:
The study is a multicenter, prospective clinical study aimed at evaluating the efficacy and safety of Huaier Granule in postoperative adjuvant treatment of resectable pancreatic cancer

DETAILED DESCRIPTION:
The study is a multicenter, prospective clinical study, expected to include subjects who visited the selected research center from April 2024 to March 2026, underwent radical tumor resection surgery, and were pathologically diagnosed with pancreatic adenocarcinoma. The subjects are divided into two groups. One group is the standard chemotherapy group, with a planned inclusion of no less than 428 subjects. The chemotherapy will be treated using the Class 1A chemotherapy regimen recommended by the 2022 version of the CSCO guidelines; One group is the Huaier treatment group, with a planned inclusion of no less than 214 subjects. All subjects voluntarily give up the postoperative adjuvant treatment recommended by the guidelines and only choose Huaier granules for postoperative adjuvant treatment. A total of no less than 642 subjects are planned to be included.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 80 years old, regardless of gender;
* Pancreatic cancer was diagnosed by histopathology after radical surgery within 12 weeks before enrollment;
* Did not receive neoadjuvant therapy before surgery and did not receive any adjuvant therapy after surgery;
* ECOG score 0-3 points;
* Those who choose to use standard chemotherapy independently based on their own situation, or choose Huaier granules for subsequent treatment, voluntarily participate in and cooperate with various research work, including but not limited to cooperating with treatment and follow-up, cooperating with researchers for data collection, and not actively taking other treatments.
* The subjects voluntarily signed a written informed consent form before participating in this study.

Exclusion Criteria:

* Known to be allergic to the components of Huaier granules or to avoid or use Huai er granules with caution (Huaier group);
* Difficulties in taking oral medication due to active gastrointestinal bleeding, perforation, gastric paralysis, etc;
* Suffering from serious mental illness or other reasons that the researcher deems unsuitable to participate in this study.
* History of merging with other malignant tumors;
* Patients with concomitant myocardial infarction, cerebral infarction, and other thromboembolic diseases requiring surgical treatment;
* Concomitant severe infection;
* Child Pugh C-grade liver function, renal function 2-5 grades (glomerular filtration rate<90ml/min);
* Pregnant or lactating women or those planning to conceive;
* The patient has received other traditional Chinese patent medicines and simple preparations with anti-tumor effect, chemotherapy or physical therapy in the past 4 weeks(including but not limited to compound cantharidin capsules, cinobufotalin capsules, Kangai injection, please refer to the drug instructions for details).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | Start of treatment until 2-year follow-up
  It is defined as the time from the first day after radical resection of pancreatic cancer to recurrence or all-cause death of pancreatic cancer.

SECONDARY OUTCOMES:
Overall survival | Start of treatment until 2-year follow-up
  It is defined as the time between the start date of enrollment and the recorded date of all-cause death. For subjects who were lost to follow-up before death, the last follow-up time is usually calculated as the time of death.
Progression-free survival | Start of treatment until 2-year follow-up
  It is defined as the time between the start date of enrollment and the date of imaging progression or all-cause death evaluated by the investigator.
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | Start of treatment until 2-year follow-up
  The definitions and severity grading of AE and SAE refer to the corresponding descriptions in the definition and evaluation section of AE. The incidence rate is defined as the proportion of patients with AE and SAE to the corresponding total population.
The incidence and severity of ADR, severe adverse reactions (SADR), suspicious and unexpected severe adverse reactions (SUSAR) | Start of treatment until 2-year follow-up
  The definitions and severity grading of ADR, severe ADR, and SUSAR refer to the corresponding descriptions in the definition and evaluation section of AE. The incidence rate is defined as the proportion of patients with ADR, severe ADR, and SUSAR to the corresponding total population.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Wang, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Zheng Wang, Xi'an, Shannxi, China